CLINICAL TRIAL: NCT00732459
Title: Clinical Trial of The Myocardial Protective Effects of Repeated Electroacupuncture Preconditioning in Heart Valve Replacement Surgery
Brief Title: Clinical Trial of Electro-Acupuncture Preconditioning in Patients Underwent Heart Valve Replacement Surgery
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Xijing Hospital (Other)
Collaborators: Air Force Military Medical University, China (Other)
Responsible Party: Lize Xiong / Director of Department of Anasthesiology of Xijing Hospital, Xijing Hospital of Fourth Military Military Medical University
Other Study IDs: XJ-20080808
Record Dates: First submitted 2008-08-09; First posted 2008-08-12 (Estimated); Last update posted 2008-08-18 (Estimated); Status verified 2008-08

CONDITIONS: Rheumatic Valve Disease
Keywords: myocardial protection; cardiac surgery; heart valve replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: electro-acupuncture preconditioning group
  Interventions: Device: Electro-acupuncture preconditioning
- 2: control group

INTERVENTIONS:
Device: Electro-acupuncture preconditioning — electro-acupuncture
  Other Names: Huatuo Brand; Type SDZ-II
  Groups: 1

SUMMARY:
The purpose of this study is to investigate the protective effect of electro-acupuncture preconditioning in patients underwent cardiac surgery.

DETAILED DESCRIPTION:
Heart valve replacement surgery has been proved to be an effective method in treating both regenerative and rheumatic valve disease. Current studies showed that cardiopulmonary bypass (CPB) and operation related myocardial injury, as indicated by the release of perioperative cardiac enzymes, is associated with worse patient morbidity and mortality after elective valve replacement surgery. Although the actual mechanism is still unclear, it has been shown that ischemic preconditioning is one potential strategy for reduction of myocardial injury in open heart surgery. Recently, Electro- acupuncture (EA) was proved to produced cerebral protective and antiarrhythmic effects by mimicking ischemic preconditioning. This study aims to assess whether electroacupuncture preconditioning is also effective in reducing myocardial injury in adults with acquired heart valve disease undergoing elective valve replacement surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients who have the indication for aortic or mitral valve replacement
* patients would like to accept the follow-up and sign the informed consent
* patients with heart function of NYHA I-III degree.

Exclusion Criteria:

* pregnant or nursing women
* comorbid with coronary artery disease
* patients with heart function of NYHA IV degree
* renal dysfunction with serum creatinine level>or=2mg/dl(177umol/L)
* anticipated life span < 12 months
* enrollment in other clinical trials at the same time not reaching the primary endpoint and probably interference the present trial.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study enrolls a group of 40-65years patients who have heart valve disease who need valve replacement.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2007-01; Primary Completion 2008-07 (Actual); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
late loss | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Lize Xiong, M.D., Study Chair — Director of Department of Anasthesiology of Xijing Hospital, Fourth Military Medical University
Locations (1):
- Department of Anesthesiology of Xijing Hospital, Fourth Military Medical University, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Yang L, Yang J, Wang Q, Chen M, Lu Z, Chen S, Xiong L. Cardioprotective effects of electroacupuncture pretreatment on patients undergoing heart valve replacement surgery: a randomized controlled trial. Ann Thorac Surg. 2010 Mar;89(3):781-6. doi: 10.1016/j.athoracsur.2009.12.003. PMID 20172127